CLINICAL TRIAL: NCT04134533
Title: Motor Functional Level and Quality of Life According to Feeding Types in Children With Cerebral Palsy
Brief Title: Comparison of Motor Functions and Quality of Life According to Feeding Type in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Emre CENGIZ, Research Assistant, Hacettepe University
Other Study IDs: Feeding Types in CP
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Feeding Group: Children with cerebral palsy who fed orally according to the Functional Oral Intake Scale
  Interventions: Other: Gross Motor Function Measurement
- Non-Oral Feeding Group: Children with cerebral palsy who fed non-orally according to the Functional Oral Intake Scale.
  Interventions: Other: Gross Motor Function Measurement

INTERVENTIONS:
Other: Gross Motor Function Measurement — These instruments will be used for determine the gross motor functional level and quality of life of the children with cerebral palsy and anxiety, depression levels of caregivers.
  Other Names: Pediatric Quality of Life Inventory; Beck Anxiety Inventory; Beck depression Inventory; Gross Motor Function Classification System

SUMMARY:
The aim of this study is to compare motor functions and quality of life of the children, and anxiety and depression levels of caregivers according to feeding type of children with cerebral palsy.

DETAILED DESCRIPTION:
The aim of this study is to compare motor functions and quality of life of the children, and anxiety and depression levels of caregivers according to feeding type of children with cerebral palsy. Children will be divided into two groups: children with oral feeding and children with non-oral feeding, according to Functional Oral Intake Scale. Gross Motor Function Classification System will be used for classify children according to gross motor function, Gross Motor Function Measurement will be used for evaluate gross motor functions, and parent-reported Pediatric Quality of Life Inventory will be used for evaluate quality of life of children. To measure caregivers' anxiety and depression levels will be assessed by using Beck Depression Inventory and Beck Anxiety Inventory. Parametric or non-parametric tests will be applied according to the variables distribution. Through this analyses, determination of the difference between feeding type groups and other categorical and continuous variables will be decided.

ELIGIBILITY:
Inclusion Criteria:

* Children who were diagnosed with CP
* Aged between 5-18 years
* Must have cooperation
* Feed by orally or non-orally

Exclusion Criteria:

* Having other accompanying neurodegenerative diseases.
* Acute respiratory tract infection
* Complications of enteral feeding

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Cerebral Palsy
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Gross motor Function Measurement | 2 months
  The Gross Motor Function Measurement (GMFM) is an observational clinical tool to evaluate motor function of children with CP. It has five basic sections that evaluate motor function in detail, including lying and rolling; sitting; crawling and kneeling; standing; and walking, running, and jumping, with a total of 88 items. Each evaluation is scored according to the level of achieving gross motor function without considering the quality of movement. While children performing each task in the GMFM, a physiotherapist scored each evaluation on a Likert scale between 0 to 3, of which 0 means 'Does not initiate' and 3 means 'Completes'.

SECONDARY OUTCOMES:
Gross Motor Function Classification System | 2 months
  The Gross Motor Function Classification System (GMFCS) was used to classify the level of gross motor functions in children with CP, and levels were based on child-initiated movement abilities, with emphasis on sitting, displacement, and mobility. The GMFCS uses a rating system of Level I to Level V, of which Level I shows the most independent functional motor level and Level V shows the most dependent functional motor level.
Pediatric Quality of Life Inventory | 2 months
  Pediatric Quality of Life Inventory (PedsQL) was used to measure the parent-reported quality of life of children. The items of the PedsQL were scored between 0 to 100, of which 100 means "never", 75 means "almost never", 50 means "sometimes", 25 means "often", and 0 means "almost always". Points are collected and divided by the number of items filled to obtain the total score. Higher scores indicate better health-related quality of life.
The Turkish version of the Beck Depression Inventory and Beck Anxiety Inventory | 2 months
  The Turkish version of the Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI) were used to measure anxiety and depression levels of caregivers of children with CP. Both scales consist of 21 question and scored between 0-3. The highest score is 63.Higher scores indicate more severe anxiety or depression of an individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No